CLINICAL TRIAL: NCT03361878
Title: Pharmacokinetics of Metformin Intolerance
Acronym: POMI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NHS Tayside (Other Government)
Collaborators: University of Southern Denmark (Other); University of Dundee (Other); Helmholtz Zentrum München (Industry)
Responsible Party: Principal Investigator, Laura McCreight, Clinical Research Fellow, NHS Tayside
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013DM06
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2; Metformin Adverse Reaction
Keywords: Metformin; Intolerance; Pharmacokinetics
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Two arms - metformin tolerant and metformin intolerant. All participants given single dose of metformin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin Tolerant (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride
- Metformin Intolerant (Active Comparator)
  Interventions: Drug: Metformin Hydrochloride

INTERVENTIONS:
Drug: Metformin Hydrochloride — Single dose of 500mg oral metformin

SUMMARY:
Pharmacokinetic study of metformin intolerance

DETAILED DESCRIPTION:
This pharmacokinetic study recruited white European individuals with type 2 diabetes, who had previously been exposed to metformin and met the criteria for tolerance or intolerance. Intolerance was defined as previous exposure to metformin (maximum of 1000mg once daily for up to 8 weeks) but discontinued treatment with patient reported or documentation of gastrointestinal upset, leading to discontinuation (Criterion 1). Alternatively, intolerance was defined as inability to increase metformin dose above 500mg without experiencing gastrointestinal side-effects, despite having an HbA1c >53mmol/mol (Criterion 2). Tolerant individuals were defined as those taking 2000mg metformin daily in divided doses, with no side effects. Ten tolerant and ten intolerant individuals were recruited.

Participants gave written consent. They attended the research centre fasted from midnight. A baseline blood test was taken before a single dose of oral metformin was administered at 0900, with further bloods taken at 11 time points over the following 24 hours. A 24 hour urine collection was completed.

Blood samples were analysed for plasma metformin, and serum lactate concentrations.

ELIGIBILITY:
Inclusion Criteria:

* White European
* Type 2 diabetes
* Meet criteria for tolerance or intolerance as described

Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) <60
* Cognitive impairment
* Pregnancy
* Concurrent treatment with: acarbose, cephalexin, cimetidine, pyrimethamine, or tyrosine kinase inhibitors
* History of gastric bypass
* Evidence of slowed gastric or intestinal motility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05-04 (Actual); Primary Completion 2016-05-05 (Actual); Study Completion 2016-05-05 (Actual)

PRIMARY OUTCOMES:
Metformin AUC | 24 hours
  Area under the metformin concentration-time curve

SECONDARY OUTCOMES:
Lactate | 24 hours
  Change in lactate concentration (incremental AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Laura McCreight, MBChB, Principal Investigator — University of Dundee

IPD SHARING:
Plan to Share IPD: Undecided
Participants have been consented for data sharing. Only anonymised data would be shared.